CLINICAL TRIAL: NCT03425097
Title: A Randomized, Double Blind, Crossover Trial Comparing Fexofenadine to Placebo for the Treatment of Proton Pump Inhibitor Refractory Gastroesophageal Reflux Symptoms
Brief Title: Fexofenadine Use in Gastroesophageal Reflux Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to insufficient evidence for Fexofenadine efficacy to treat GERD symptoms after the interim analysis.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Zikos, Fellow in Gastroenterology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-44650
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — fexofenadine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fexofenadine then Placebo (Experimental): Patients in this group will get 2 weeks of fexofenadine, then 1 week of nothing, then 2 weeks of placebo.
  Interventions: Drug: Fexofenadine; Drug: Placebo - Cap
- Placebo then Fexofenadine (Experimental): Patients in this group will get 2 weeks of placebo, then 1 week of nothing, then 2 weeks of fexofenadine.
  Interventions: Drug: Fexofenadine; Drug: Placebo - Cap

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine 180 mg in the morning
Drug: Placebo - Cap — Placebo cap in the morning

SUMMARY:
The investigators wish to study the effectiveness of Fexofenadine (an over the counter allergy pill) for the treatment of gastroesophageal reflux symptoms in patients who still have symptoms despite being on a proton pump inhibitor. The investigators will do this by giving participants both Fexofenadine (an H1 blocker) for 2 weeks and placebo (sugar pill) for 2 weeks. The participants will not know which drug they are getting at a particular time. This will help the investigators better assess the true effectiveness of Fexofenadine.

DETAILED DESCRIPTION:
Around 18-28% of North American adults have gastroesophageal reflux symptoms once per week. Of those patients up to 60% may have an inadequate response to proton pump inhibitors and have persistent symptoms. One possible explanation is that this group of patients has nerve related pain. It is thought that H1 receptor activation may sensitize the gastrointestinal tract and esophagus to pain. H1 blockers such as anti-histamines may play a role in treatment of gastroesophageal reflux symptoms that are refractory to proton pump inhibitors by reducing pain perception. The investigators wish to conduct a randomized control trial to test this hypothesis. The investigators will do this by giving participants both Fexofenadine (an H1 blocker) for 2 weeks and placebo (sugar pill) for 2 weeks. The participants will not know which drug they are getting at a particular time. This will help the investigators better assess the true effectiveness of Fexofenadine.

ELIGIBILITY:
Inclusion Criteria:

* A minimum 6-month history of heartburn and regurgitation, as their main symptom
* Experience at least 3-4 days with episodes of heartburn or regurgitation per week
* Female patients who are postmenopausal or using acceptable methods of birth control.

Exclusion Criteria (selected)

* Esophageal stricture
* Primary esophageal motility disorder
* Systemic sclerosis
* Active inflammatory bowel disease
* Zollinger-Ellison syndrome
* Active gastric or duodenal ulcer
* Active infectious or inflammatory conditions of the small or large intestine
* Malabsorption syndromes of the intestine
* History of gastrointestinal cancer
* Current active cancer
* Prior gastric or intestinal surgery
* Pregnant or breast feeding
* Other serious psychiatric or medical disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants entered a 7 day run in period prior to randomization.
Groups:
- Fexofenadine Then Placebo: Patients in this group will get 2 weeks of fexofenadine (180 mg), then 1 week of nothing, then 2 weeks of placebo.
- Placebo Then Fexofenadine: Patients in this group will get 2 weeks of placebo, then 1 week of nothing, then 2 weeks of fexofenadine (180 mg)
Period: Treatment Period 1 (2 Weeks)
Arm/Group | Fexofenadine Then Placebo | Placebo Then Fexofenadine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout Period (1 Week)
Arm/Group | Fexofenadine Then Placebo | Placebo Then Fexofenadine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Treatment Period (2 Weeks)
Arm/Group | Fexofenadine Then Placebo | Placebo Then Fexofenadine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Patients in this group will get 2 weeks of fexofenadine (180 mg) or matching placebo, then 1 week of nothing, then 2 weeks of the opposite treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants] — Population: Age data are available for only 6 participants
  Participants
    40-49 years: number analyzed (Participants) | 6
    40-49 years | 1
    50-59 years: number analyzed (Participants) | 6
    50-59 years | 1
    60-69 years: number analyzed (Participants) | 6
    60-69 years | 2
    70-79 years: number analyzed (Participants) | 6
    70-79 years | 1
    80-89 years: number analyzed (Participants) | 6
    80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data are available for only 9 participants
  Participants
    number analyzed (Participants) | 9
    Female | 2
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data are available for only 9 participants
  Participants
    number analyzed (Participants) | 9
    Hispanic or Latino | 0
    Not Hispanic or Latino | 9
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Days With Reflux
Time Frame: 2 weeks per treatment
Population: Participants with available data are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of days
Groups:
- Run-in Period: Participants entered a 1 week run-in period prior to randomization.
- Fexofenadine: Fexofenadine (180 mg) for 2 weeks
- Placebo: Fexofenadine placebo for 2 weeks
Arm/Group | Run-in Period | Fexofenadine | Placebo
Number analyzed (Participants) | 6 | 6 | 6
percentage of days | 83.4 [59.4 to 107.4] | 52.4 [4.3 to 100.4] | 52.4 [12.5 to 92.2]

2. Primary Outcome: Mean Number of Reflux Episodes Per Day
Time Frame: 2 weeks per treatment
Population: Participants with available data are included in the analysis
Measure: Mean (95% Confidence Interval); unit: episodes
Arm/Group | Run-in Period | Fexofenadine | Placebo
Number analyzed (Participants) | 6 | 6 | 6
episodes | 1.74 [0.73 to 2.75] | 0.69 [-0.01 to 1.40] | 0.67 [-0.05 to 1.29]

3. Primary Outcome: Mean GERD-HRQL Questionnaire Score
Description: The questionnaire consists of 10 questions with responses of 0-5. The responses of the 10 questions are totaled (range of 0-50) where a higher total indicates more severe disease than a lower total.
Time Frame: 2 weeks per treatment
Population: Participants with available data are included in the analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Run-in Period | Fexofenadine | Placebo
Number analyzed (Participants) | 6 | 6 | 6
score on a scale | 16.2 [2.5 to 29.8] | 9.8 [-1.5 to 21.2] | 12.3 [4.0 to 20.7]

4. Primary Outcome: Mean Symptom Severity Score
Description: Severity of reflux symptoms on a scale of 0-4 (0=none, 1=mild, 2=moderate, 3=severe, 4=very severe)
Time Frame: 2 weeks per treatment
Population: Participants with available data are included in the analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Run-in Period | Fexofenadine | Placebo
Number analyzed (Participants) | 6 | 6 | 6
score on a scale | 1.2 [0.6 to 1.9] | 0.8 [-0.03 to 1.5] | 0.7 [-0.02 to 1.4]

5. Primary Outcome: Mean Rescue Medications Per Day
Description: Medications such as Tums or Pepcid can be used if reflux symptoms are severe and relief is needed (additional doses of proton pump inhibitors are not allowed beyond the regular dosing)
Time Frame: 2 weeks per treatment
Population: Participants with available data are included in the analysis
Measure: Mean (95% Confidence Interval); unit: medications
Arm/Group | Run-in Period | Fexofenadine | Placebo
Number analyzed (Participants) | 6 | 6 | 6
medications | 0.29 [-0.31 to 0.89] | 0.52 [-0.75 to 1.80] | 0.17 [-0.14 to 0.47]

6. Secondary Outcome: Patient Medication Preference
Description: Patients will be asked which medication they think better helps treat their reflux symptoms, placebo or Fexofenadine.
Time Frame: Will be assessed at the end of the trial (total trial time is 6 weeks)
Population: Data were not collected for this outcome measure
Arm/Group | Run-in Period | Fexofenadine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Count of Participants With Side Effects
Description: Patients will write down side effects at the end of each treatment period. If severe patients should seek medical attention immediately and report the side effects to us.
Time Frame: Will be assessed at the end of the initial treatment period (2 weeks) and at the end of the crossover period (2 weeks)
Population: Participants with available data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Fexofenadine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fexofenadine (N=11) | Placebo (N=11)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was underpowered as it did not meet its planned sample size of 40 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03425097/Prot_SAP_000.pdf